CLINICAL TRIAL: NCT05743348
Title: COVID-19 e Telepsychotherapy: Which Variables Affect Therapeutic Experience?
Acronym: TELECOVID
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 23C123
Record Dates: First submitted 2023-02-22; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Telepsychotherapy
MeSH Terms: interventions — Mental Health Teletherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Telepsychotherapy — Remotely delivered psychotherapy sessions

SUMMARY:
COVID-19 pandemic forced a widespread adoption of telemedicine, including telepsychotherapy.

Telepsychotherapy has been proven to be effective before COVID-19 breakout (Poletti et al., 2020); however, both patients and therapists were skeptical about this modality.

The aim of this study is to probe the experience of telepsychotherapy in both patients and therapists, during the COVID-19 lockdown. Thus, when the adoption of online colloquia was mandatory and not an option.

Crucially, studying the experience of telepsychotherapy during the COVID-19 pandemic allows i) investigating also the experience of those patients and therapists that were not favorable to this kind of intervention and ii) comparing the experience of therapy in the online and face-to-face modality, in the same patients and therapists. Furthermore, we collect several psychological variables that possibly influence the experience and efficacy of telepsychotherapy (e.g., personality traits, attachment state of mind, previous traumatic experiences) to define the psychological profile behind a favorable or negative experience of telemedicine in both patients and therapists. As crucial novelty, this information is collected in both patients and their therapists, allowing the direct comparisons between the experience of the therapeutic relationship (e.g., empathy, alliance) from two different point of views.

The results of the present study may help in the definition of possible subgroups of patients who may be sufficiently responsive to telepsychotherapy and those who may benefit - exclusively - of face-to-face interventions.

ELIGIBILITY:
Inclusion Criteria:

* Licensed and currently practicing psychotherapists
* Individuals currently undergoing a psychotherapy

Exclusion Criteria:

* not applicable

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study addresses both licensed and currently practicing psychotherapists and their patients, namely individuals currently undergoing a psychotherapy
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Telepsychotherapy perception | At enrollment
  Psychometric measures of general perception/experience on the remotely delivered psychotherapy as far as efficacy and interpersonal factors are concerned

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No